CLINICAL TRIAL: NCT00840775
Title: Clinical Protocol Presillion™ and Presillion™ Plus Stent Systems
Brief Title: PIONIR Study (Presillion™ and Presillion™ Plus Stent Systems)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medinol Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CV103-01
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Ischemic Heart Disease
Keywords: Stent; interventional cardiology; catheterization; symptomatic ischemic heart disease
MeSH Terms: conditions — Myocardial Ischemia | interventions — Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Presillion™ Stent System (Other)
  Interventions: Device: Catheterization, stent deployment

INTERVENTIONS:
Device: Catheterization, stent deployment — Standard catheterization procedure including Bare Metal Stent deployment.
  Other Names: CoCr Coronary Stent; Coronary Stent

SUMMARY:
The purpose of this study is to collect and analyze additional information about the safety and effectiveness of the Presillion™ Stent System in the treatment of de novo stenotic lesions in native coronary arteries.

DETAILED DESCRIPTION:
This is a post market, non-randomized, multi-center, prospective, single arm clinical study that will be conducted at up to 25 sites in Europe and Israel. All patients will be followed at 30 days, 6 months, 9 months and 1 year post index stenting procedure.

The primary endpoint will be the incidence of target vessel failure (TVF, see definition below) within 270 days of treatment with the Presillion™ Stent System. This rate will be compared with a performance goal derived using a meta-analysis of the standard-of-care therapy, coronary stenting with bare metal stents. This data will be used to support the PMA application for the Presillion™ Stent System.

ELIGIBILITY:
Inclusion Criteria:

1. Patient >= 18 years old.
2. Eligible for Percutaneous Coronary Intervention (PCI).
3. Patient understands the nature of the procedure and provides written informed consent prior to the catheterization procedure.
4. Patient is willing to comply with specified follow-up evaluation and can be contacted by telephone.
5. Acceptable candidate for coronary artery bypass graft (CABG) surgery.
6. Stable angina pectoris (Canadian Cardiovascular Society (CCS) 1, 2, 3 or 4) or unstable angina pectoris (Braunwald Class 1-3, B-C) or a positive functional ischemia study (e.g., ETT, SPECT, Stress echocardiography or Cardiac CT).
7. Male or non-pregnant female patient (Note: females of child bearing potential must have a negative pregnancy test prior to enrollment in the study).

Exclusion Criteria:

1. Currently enrolled in another investigational device or drug trial that has not completed the primary endpoint or that clinically interferes with the current study endpoints.
2. Previously enrolled in another stent trial in the previous 2 years.
3. ANY planned elective surgery or percutaneous intervention within subsequent 9 months.
4. A previous coronary interventional procedure of any kind within the 30 days prior to the procedure.
5. The subject requires staged procedure of either the target or any non-target vessel within 9 months post-procedure.
6. Previous drug eluting stent (DES) deployment anywhere in the target vessel.
7. Any drug eluting stent (DES) deployment anywhere within the past 12 months
8. Co-morbid condition(s) that could limit the patient's ability to participate in the trial or to comply with follow-up requirements, or impact the scientific integrity of the trial.
9. Concurrent medical condition with a life expectancy of less than 12 months.
10. Known hypersensitivity or contraindication to aspirin, heparin or bivalirudin, clopidogrel or ticlopidine, cobalt, nickel, L-605 Cobalt chromium alloy or sensitivity to contrast media, which cannot be adequately pre-medicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2009-04; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Target vessel failure (TVF) | 270 days

CONTACTS AND LOCATIONS:
Locations (16):
- Belgium (4):
  - ZNA Middelheim, Antwerp
  - UZ Brussel, Brussels
  - CHU Charleroi, Charleroi
  - CHU de Liege, Liège
- Germany (6):
  - Herz-Kreislauf-Zentrum Segeberger Kliniken, Bad Segeberg
  - Charité - Campus Benjamin Franklin, Berlin
  - CardioVascular Center Frankfurt Sankt Katharinen, Frankfurt
  - University Hospital of Heidelberg, Heidelberg
  - Helios Klinkum, Siegburg
  - Schwarzwald-Baar Klinikum Villingen-Schwenningen GmbH, Villingen-Schwenningen
- Israel (4):
  - EMEK Medical Center, Afula
  - Hadassah Medical Organization, Jerusalem
  - Sanz Medical Center, Laniado Hospital, Netanya
  - Assaf Harofeh Medical Center, Ẕerifin
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Lund University Hospital, Lund

REFERENCES:
- See also: Related Info — http://medinol.com